CLINICAL TRIAL: NCT00182416
Title: Second Canadian Trial of Physiologic Pacing (CTOPP II): Pilot Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Medtronic (Industry); Sunnybrook Health Sciences Centre (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTMG-2005-CTOPPII
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Pacemaker Dependence
Keywords: pacemakers; atrial fibrillation; stroke; cardiovascular death
MeSH Terms: conditions — Atrial Fibrillation; Stroke

INTERVENTIONS:
Device: pacemaker

SUMMARY:
Pacemaker therapy has been recognized as effective for the control of sinus and atrio-ventricular (AV) node dysfunction. Single chamber pacing when compared with dual chamber pacing, has numerous advantages of low complication rates, lower cost, better longevity, with non-inferiority in the quality of life and hard outcomes proven in direct randomized comparisons. However, comparison between single and dual chamber pacers was never adequate, since not more then half of the patients in the trials were actually using pacemakers for the majority of the time. Routine dual chamber pacing using a right ventricle apical lead is also associated with significant increase in peri-operative and remote complications. Some of these complications may be related to ventricular desynchronization secondary to the pacing location, which is potentially avoidable by using biventricular pacing. A randomized trial which will compare single chamber rate responsive pacing to the best available modification of dual chamber pacing (biventricular pacing) in suitable patients is therefore warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic bradycardia and is a candidate for first pacemaker implantation
* Patient has high risk of being pacemaker dependent by (at least one of the following):

  1. Average heart rate of 60 or less on pre-implant Holter
  2. Maximal heart rate of 60 in patient on telemetry monitoring 12 hrs preoperatively, when not under medications decreasing heart rate, or under chronic medical treatment inducing bradycardia, which is unlikely to be changed
  3. First degree AV block with PR intervals > 300 ms, or second degree AV block at heart rates <= 80 bpm.
  4. Dependence for 12 hrs when on temporary pacemaker set at 50 bpm if bradycardia is not secondary to medication, or under chronic medical treatment inducing bradycardia, which is unlikely to be changed.

Exclusion Criteria:

* Age <= 65 years
* Chronic Atrial Fibrillation
* Indication for ICD
* Non-cardiovascular death is likely to occur within 3 years
* Geographical, social, or psychiatric reasons making follow-up problematic

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300
Dates: Start 2004-05; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Predictors of future pacemaker dependence
Feasibility of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Crystal, MD, Study Chair — Sunnybrook & Women's College Health Sciences Centre; Robin S Roberts, Principal Investigator — McMaster Univeristy, Department of Clinical Epidemiology & Biostatistics; Stuart Connolly, MD, Principal Investigator — Hamilton Health Sciences - General Division; Paul Dorian, MD, Principal Investigator — Unity Health Toronto
Locations (5):
- Canada (5):
  - Hamilton Health Sciences - General Division, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario